CLINICAL TRIAL: NCT02030743
Title: A Study of Visual Attention Training to Improve Balance and Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: King Saud University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19456
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2015-12

CONDITIONS: Accidental Falls
Keywords: Falls; Older adults; Balance; Mobility; Visual attention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visual training (Active Comparator): Training in visual attention
  Interventions: Other: Visual training
- Usual activity (Placebo Comparator): Usual activity
  Interventions: Other: Visual training

INTERVENTIONS:
Other: Visual training — 6 training sessions with computerised visual attention paradigm

SUMMARY:
The purpose of this study is to determine if training visual attention improves balance and mobility, and reduces falls in older adults.

DETAILED DESCRIPTION:
Visual training in visual attention is compared with activity as usual.

ELIGIBILITY:
Inclusion Criteria:

* healthy older adults
* Visual acuity 6/12 or better
* able to speak English

Exclusion Criteria:

* No known dementia or cognitive impairment
* not dependent on a walker or cane

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Balance on force plate platform | after 4 weeks
  Standard deviation of the medial lateral (ML) and anterior posterior (AP) center of pressure, ML and AP CoP maximum sway, ML and AP CoP range in each direction (range = maximum excursion - minimum excursion) and the cumulative path length in cms

SECONDARY OUTCOMES:
Mini-BESTest (Balance evaluation) | after 4 weeks
  14 short balance tests divided under four domains of balance control; 1) anticipatory body control, 2) reactive postural control, 3) sensory orientation and 4) balance during dynamic gait

OTHER OUTCOMES:
One Legged Stance Test | after 4 weeks
  The duration participant is able to maintain their balance on one leg up to 30 seconds is recorded
Sit to Stand test | after 4 weeks
  Participant is timed for 5 sit to stands
Timed Up and Go test | after 4 weeks
  the TUG alone and the TUG with a cognitive task (TUGco)
5 Metre Walking test | after 4 weeks
  Time taken to walk 5m in a straight line with no obstacles.

CONTACTS AND LOCATIONS:
Overall Officials: Susan J. Leat, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada